CLINICAL TRIAL: NCT05864755
Title: Hepatic Arterial Infusion Chemotherapy (HAIC) Plus Tremelimumab, Durvalumab and Bevacizumab as Conversion Therapy for Potentially Resectable Hepatocellular Carcinoma (HCC): a Single Center, Open Label, Single Arm, Phase II Trial
Brief Title: HAIC Combined With Durvalumab, Tremelimumab and Bevacizumab as Conversion Therapy for Potentially Resectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L20230427
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-05

CONDITIONS: Unrescetable Hepatocellular Carcinoma
Keywords: Unrescetable Hepatocellular Carcinoma; Durvalumab; Tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC+Durvalumab+Tremelimumab+Bevacizumab (Experimental)
  Interventions: Drug: HAIC+Durvalumab+Tremelimumab+Bevacizumab

INTERVENTIONS:
Drug: HAIC+Durvalumab+Tremelimumab+Bevacizumab — Tremelimumab：300mg, only once in cycle 1.Durvalumab: 1500mg, iv,q3w Bevacizumab: 15mg/kg, iv, q3w HAIC: Oxaliplatin plus Fluorouracil/Leucovorin

SUMMARY:
To evaluate the efficacy and safety of HAIC combined with Durvalumab, Tremelimumab and Bevacizumab as first-line therapy in Unresectable hepatocellular carcinoma

DETAILED DESCRIPTION:
An open label, single-arm, single center, phase II study evaluating HAIC combined with Durvalumab, Tremelimumab and Bevacizumab as first-line therapy in unresectable hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Provide a written informed consent form (ICF) signed and dated by the patient/legal representative before conducting any research specific procedures, sampling, and analysis specified in the protocol.
2. Before collecting genetic analysis samples (optional), provide a signed and dated written informed consent form for genetic research.
3. At the time of screening, the age should be ≥ 18 years old. For patients under the age of 20 who are enrolled in China, written informed consent from the patient and their legal representative should be obtained.
4. Based on the histopathology results of tumor tissue, a patient with stage C hepatocellular carcinoma complicated with portal vein tumor thrombus BCLC was diagnosed, with portal vein tumor thrombus type I to III. (Cheng's classification indicates that the tumor thrombus is mainly located at the level of the liver segment (secondary branch of the portal vein); Type II refers to the spread of cancer thrombi invading the left or right branch of the portal vein (primary branch of the portal vein); Type III refers to cancer thrombus invading the main portal vein; Type IV refers to tumor thrombus invading superior mesenteric vein or inferior vena cava.
5. No evidence of extrahepatic diseases was found in baseline chest/abdominal/pelvic imaging
6. The disease is not suitable for radical surgery, transplantation, or radical ablation
7. The disease must be suitable for TACE and HAIC treatment, and it is expected that TACE treatment for local lesions will not exceed 4 times within 16 weeks [DEB-TACE]
8. The Child Pugh grading of liver function is Grade A,the Eastern Oncology Collaborative Group (ECOG) physical fitness score was 0 or 1
9. Patients with HBV infection [showing positive hepatitis B B virus surface antigen (HBsAg), and/or positive hepatitis B core antibody (anti HBcAb)] and detectable HBV DNA (≥ 10IU/mL or higher than the detection limit according to the local experimental standard) must receive antiviral treatment according to the institutional diagnosis and treatment routine to ensure adequate virus suppression (HBV DNA ≤ 2000IU/mL) before enrollment. Patients must maintain antiviral treatment during the study period and within 6 months after the last administration of the study drug. For patients who are positive for hepatitis B core antibody (HBc) but have not detected HBV DNA (<10 IU/ml or below the detection limit of local laboratory standards), antiviral treatment is not required before enrollment. These patients need to monitor HBV DNA levels during each course of treatment, and once HBV DNA is tested (≥ 10 IU/mL or below the detection limit of local laboratory standards), antiviral treatment begins. Patients who can detect HBV DNA must begin and maintain antiviral therapy during the study period and within 6 months after the last administration of the study drug.
10. According to the following mRECIST criteria, at least one measurable intrahepatic lesion is suitable for repeated evaluation: in intravenous contrast-enhanced CT or MRI scans, the liver lesion shows typical features of HCC, namely arterial phase vascular enhancement, venous phase or delayed phase enhancement rapidly disappears in the non necrotic part at baseline (arterial phase IV contrast agent enhancement), and its longest diameter can be accurately measured to be ≥ 10 mm
11. The definition of good organ and bone marrow function is as follows. Within 14 days before the start of the first dose, standards "a", "b", "c", and "f" cannot be met through blood transfusion, infusion, or receiving supportive therapies such as growth factors

    1. Hemoglobin ≥ 9.0 g/dL
    2. Absolute neutrophil count ≥ 1000/µ L
    3. Platelet count ≥ 75000/ μ L
    4. Total bilirubin ≤ 2.0 × Upper limit of normal value (ULN)
    5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN
    6. Albumin ≥ 2.8 g/dL
    7. International normalized ratio (INR) ≤ 1.6
    8. 2+or lower urine test strip reading
    9. Calculate creatinine clearance rate (CL) ≥ 30mL/min, and measure male creatinine CL=weight (kg) using Cockcroft Fault (using actual body weight) or 24-hour urine creatinine CL × (140 Age) (mL/min) 72 × Serum creatinine (mg/dL) Female: creatinine CL=weight (kg) × (140- Age) × 0.85（mL/min）72 × Serum creatinine (mg/dL)
12. Must have an expected lifespan of at least 12 weeks
13. Weight>30 kg
14. No gender limit

Exclusion Criteria:

1. History of kidney disease or nephrotic syndrome
2. Cardiovascular diseases with clinical significance
3. Major traumatic injury occurred within the first 4 weeks of randomization
4. Known genetic factors for bleeding or thrombosis; Any previous or current evidence indicating a tendency to bleed
5. Systematic anticoagulant therapy is allowed, except for vitamin K antagonists
6. History of arterial embolism events, including stroke or myocardial infarction
7. Patients with unhealed wounds, active ulcers, or fractures. For granulation wounds in the second stage of healing, as long as there is no evidence of surface cracking or infection in patients, they meet the inclusion criteria but require wound examination every 3 weeks
8. Abdominal wall fistula or gastrointestinal perforation, refractory unhealed gastric ulcer, or active gastrointestinal bleeding within 6 months before enrollment
9. Patients who have undergone any surgery within the past 28 days (diagnostic biopsy is acceptable)
10. Uncontrolled hypertension is defined as systolic blood pressure>150 mmHg or diastolic blood pressure>90 mmHg, with or without taking antihypertensive drugs. Patients who experience an increase in blood pressure (BP) for the first time can be enrolled if using or adjusting antihypertensive drugs can lower their blood pressure to the inclusion criteria.
11. Diagnosed fibrolaminar HCC, sarcomatous HCC, or mixed cholangiocarcinoma and HCC
12. Have a history of hepatic encephalopathy within the past 12 months, or require medication to prevent or control encephalopathy (such as using lactulose, rifaximin, etc. for hepatic encephalopathy).
13. Large portal vein thrombosis was seen in the baseline/qualification test imaging, and patients with type IV procedures were excluded
14. Patients with infiltrative HCC
15. Have a history of homologous organ transplantation
16. Active or previously recorded autoimmune diseases or inflammatory diseases (including inflammatory bowel disease [such as colitis or Krohn's disease], diverticulitis [except diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome or Wegener's syndrome [such as granulomatous vasculitis, Gray's disease, rheumatoid arthritis, hypophysitis and uveitis]). There are the following exceptions to this standard:

    * Patients with vitiligo or hair loss
    * Patients with stable hypothyroidism after receiving hormone replacement therapy (such as after Hashimoto's thyroiditis) Any chronic skin disease patient who does not require systemic treatment
    * Patients with no active diseases within the past 5 years can be included, but only after consulting the research doctor can they be included Patients with celiac disease who can be controlled solely by diet
17. Uncontrolled complications, including but not limited to: persistent or active infection (except for the above HBV or HCV), symptomatic congestive heart failure, uncontrollable diabetes, uncontrollable hypertension, unstable angina pectoris, uncontrollable arrhythmia, active ILD, severe chronic GI disease with diarrhea, or suffering from a condition that may limit compliance with the study requirements Mental illness/social issue conditions that significantly increase the risk of AE or affect the subject's ability to provide written informed consent.
18. History of other primary malignant tumors, except for the following situations Malignant tumors that have been treated for the purpose of cure, and have no known active diseases for ≥ 5 years before the first administration of IP, with a low potential risk of recurrence

    - Fully treated non melanoma skin cancer or malignant lentiginous nevus without disease evidence Fully treated in situ cancer with no evidence of disease
19. History of meningeal cancer
20. History of active primary immunodeficiency
21. Active infection, including tuberculosis (clinical evaluation, including clinical history, physical examination and imaging examination results, as well as tuberculosis testing according to local clinical standards) or human immunodeficiency virus (HIV 1/2 antibody positive)
22. Patients who are co infected with HBV and HCV, or co infected with HBV and hepatitis D virus (HDV). (HBV infection refers to the presence of HBsAg and/or anti HBcAb, and detectable HBV DNA ≥ 10 IU/mL or according to local laboratory standards detection limit; HCV positive infection refers to detectable HCV RNA; HDV positive infection refers to the presence of anti HDV antibodies.)
23. Except for hair loss, vitiligo, and laboratory values specified in the inclusion criteria, any unrelieved NCI (National Cancer Institute) CTCAE v5.0 ≥ Level 2 events caused by previous anti-cancer treatment
24. Known to cause allergic or hypersensitive reactions to any investigational drug or any of its excipients
25. Have a history of allogeneic bone marrow transplantation and active chronic graft versus host disease
26. Have received anti PD-1, anti PD-L1, or anti CTLA-4 treatment before the first administration of IP
27. Previously received TACE (transcatheter arterial chemoembolization), TAE (transcatheter arterial embolization), or TARE (transcatheter arterial radioembolization)
28. Previously received systemic anti-cancer treatment for HCC
29. IP has been vaccinated with attenuated live vaccine within 30 days before the first administration. Note: If enrolled, patients are not allowed to receive attenuated live vaccines during IP treatment and within 30 days after the last administration of IP.
30. Currently in use or using immunosuppressive drugs within 14 days before the first dose of IP administration. This standard has the following exceptions:

    - Intranasal, inhalation, topical steroids, or local injection of steroids (such as intra-articular injection) Whole body corticosteroid therapy with no more than 10 mg/day prednisone or its equivalent physiological dose as a preventive use of steroid hormones for hypersensitivity reactions (such as CT scan pre-treatment medication)
31. Previously received IP allocation in this study
32. Simultaneously enroll in another clinical study, unless the study is an observational (non intervention) clinical study or during the follow-up period of an intervention study
33. Prior to randomization or treatment, participants had previously participated in clinical studies of immune checkpoint inhibitors, regardless of treatment group allocation.
34. From screening to 6 months after the last administration of IP, pregnant or lactating female patients, or male or female patients with fertility, are unwilling to use efficient contraceptive measures. According to the patient's preferred and habitual lifestyle, abstinence during treatment and abstinence is an acceptable contraceptive measure.
35. Patients who, in the judgment of the researcher, are unlikely to comply with the research steps, limitations, and requirements shall not participate in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate ( ORR) per RECIST 1.1 | Up to 1 year
  Defined as proportion of patients who have a best response of CR or PR

SECONDARY OUTCOMES:
Overall survival (OS) | Up to two years
  Defined as the time from enrollment to death from any cause
Progress Free Survival (PFS) | Up to two years
  Defined as the time from enrollment to disease progression or death (whichever occurs first)
Disease Control Rate (DCR) per RECIST 1.1 | Up to one year
  Defined as proportion of patients who have CR or PR or SD
Duration of Response(DoR) per RECIST 1.1 | Up to two years
  The time from the first assessment of the tumor as CR or PR to the second assessment as PD (Progressive Disease) or death from any cause
Time To Progress(TTP) per RECIST 1.1 | Up to two years
  The time from the beginning to the first objective progression of the tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No